CLINICAL TRIAL: NCT01610453
Title: Prediction of Mode of Delivery With Transperineal Ultrasound in Women With Prolonged First Stage of Labour. A Multicentre Study
Brief Title: Prediction of Delivery With Transperineal Ultrasound in Women With Prolonged Labour. Multicentre Study
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Norwegian University of Science and Technology (Other); Haukeland University Hospital (Other); Skane University Hospital (Other); Hvidovre University Hospital (Other); Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: REK2011/731; susID155 (Registry Identifier: Stavanger University Hospital)
Record Dates: First submitted 2012-02-10; First posted 2012-06-04 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Failed Labor
Keywords: prolonged labor; cesarean section; duration of labor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ultrasound: primiparous women with prolonged labours will be eligible for examination
  Interventions: Procedure: ultrasound examination

INTERVENTIONS:
Procedure: ultrasound examination — transabdominal and transperineal ultrasound examinations

SUMMARY:
Objectives

1. To assess if head-perineum distance and angle of progression measured with transperineal ultrasound by the obstetrician on call can predict delivery mode in primiparous women with prolonged first stage of labour.
2. To compare ultrasound assessments and clinical examinations.

DETAILED DESCRIPTION:
Variables Digitally assessed cervical dilatation, fetal station and position Ultrasound measured fetal head-perineum distance. Ultrasound measured angle of progression Ultrasound assessed position

Possible confounders Ethnicity, maternal age, gestational age, BMI, induction of labour, augmentation, epidural analgesia, birth weight, head circumference

A two-dimensional ultrasound measurement will be obtained with the ultrasound device available in the delivery department. Fetal head descent is measured as the shortest distance between the outer bony limit of the fetal skull and the perineum with a curved transabdominal transducer placed transperineally between the labia in a transverse view (1).

The fetal descent will also be assessed measuring "angle of progression" as suggested by Barbera et al. The ultrasound transducer will be placed on the perineum in a mid-sagittal position between the labia below the pubic symphysis. The angle between a line through the symphysis and a line from the posterior part of the symphysis tangentially to the fetal skull contour will be measured (2)

A transabdominal scan will also be performed determining the fetal position as described previously. Positions ≥ 02.30 and ≤ 03.30 hours should be recorded as left occiput transverse and positions ≥ 08.30 and ≤ 09.30 as right occiput transverse. Positions > 03.30 and <08.30 should be recorded as occiput posterior and positions > 09.30 and < 02.30 as occiput anterior.(3).

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women with single pregnancies and gestation age > 37 weeks and prolonged first stage of labor

Exclusion Criteria:

* High risk pregnancies,
* premature deliveries,
* multiple pregnancies

Ages: 15 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: primiparous women in labor
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torbjørn M Eggebø, PhD, Principal Investigator — Helse Stavanger HF
Locations (6):
- Hvidovre Hospital, Copenhagen, Hvidovre, Denmark
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Stavanger University Hospital, Stavanger
  - St.Olavs Hospital, Trondheim
- Skåne University Hospital, Malmo, Sweden
- Addenbrooke's Hospital, Cambridge, United Kingdom

REFERENCES:
- [Background] Torkildsen EA, Salvesen KA, Eggebo TM. Prediction of delivery mode with transperineal ultrasound in women with prolonged first stage of labor. Ultrasound Obstet Gynecol. 2011 Jun;37(6):702-8. doi: 10.1002/uog.8951. Epub 2011 May 3. PMID 21308837
- [Background] Barbera AF, Pombar X, Perugino G, Lezotte DC, Hobbins JC. A new method to assess fetal head descent in labor with transperineal ultrasound. Ultrasound Obstet Gynecol. 2009 Mar;33(3):313-9. doi: 10.1002/uog.6329. PMID 19248000
- [Background] Akmal S, Tsoi E, Kametas N, Howard R, Nicolaides KH. Intrapartum sonography to determine fetal head position. J Matern Fetal Neonatal Med. 2002 Sep;12(3):172-7. doi: 10.1080/jmf.12.3.172.177. PMID 12530614
- [Result] Eggebo TM, Hassan WA, Salvesen KA, Lindtjorn E, Lees CC. Sonographic prediction of vaginal delivery in prolonged labor: a two-center study. Ultrasound Obstet Gynecol. 2014 Feb;43(2):195-201. doi: 10.1002/uog.13210. Epub 2013 Dec 22. PMID 24105705
- [Result] Eggebo TM, Hassan WA, Salvesen KA, Torkildsen EA, Ostborg TB, Lees CC. Prediction of delivery mode by ultrasound-assessed fetal position in nulliparous women with prolonged first stage of labor. Ultrasound Obstet Gynecol. 2015 Nov;46(5):606-10. doi: 10.1002/uog.14773. Epub 2015 Sep 28. PMID 25536955

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from 1. January 2012 until 30. April 2013
Groups:
- Results From Transperineal Scan: Primiparous women with prolonged labours was eligible for the study. Addenbrooke's Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge, UK and Department of Obstetrics and Gynecology, Stavanger University Hospital, Stavanger, Norway participated.
  Ultrasound examination: a transperineal sonography was done when prolonged labor was diagnosed. Prolonged labor was diagnosed in accordance with WHO recommendations in Stavanger and in accordance with NICE guidelines in Cambridge
Period: Overall Study
Arm/Group | Results From Transperineal Scan
Started | 150
Completed | 150
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Transperineal Ultrasound: Fetal head descent was assessed using a transperineal scan
Arm/Group | Transperineal Ultrasound
Number analyzed (Participants) | 150
Age, Continuous [Median (Full Range); unit: years] | 29 [18 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 0
Region of Enrollment [Number; unit: participants]
  Norway | 87
  United Kingdom | 63

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Women With Vaginal Deliveries
Description: Women were categorized in accordance to fetal descent measured by ultrasound. Head-perineum distance (HPD) ≤40 mm and angle of progression (AoP) ≥110 degrees were used as cut-off level. HPD was obtained in all 150 cases and AoP was successfully obtained in 145 cases.
Time Frame: active labor
Population: AoP could not be measured in 5 cases because only a part of the symphysis was visualized.
Measure: Number (95% Confidence Interval); unit: percentage of participants in each group
Arm/Group | Transperineal Ultrasound
Number analyzed (Participants) | 150
percentage of participants in each group
  Vaginal deliveries if HPD was ≤40 mm (n=84) | 92 [84 to 96]
  Vaginal deliveries if HPD was >40 mm (n=66) | 52 [40 to 63]
  Vaginal deliveries if AoP was ≥110 degrees (n=84) | 88 [79 to 93]
  Vaginal deliveries if AoP was <110 degrees (n=61) | 57 [45 to 69]
Statistical Analysis 1: Comparison: Transperineal Ultrasound; Women were categorized in accordance to fetal descent measured by ultrasound. Head-perineum distance ≤40 mm was used as cut-off level. Vaginal delivery was the primary outcome measure; Test type: Superiority or Other; p < 0.01, Chi-squared — A sample size calculation with alpha 0.05, power 0.8, and cut-off level of HPD at 40 mm. 146 women should be included. The calculation was based from a previous study, in which 93% with HPD ≤40 mm and 57% of with HPD > 40 mm delivered vaginally

2. Secondary Outcome: Percentage of Women With Cesarean Section
Description: The percentage of women with cesarean section was compared in cases with occiput posterior position and cases with non occiput posterior position assessed with transabdominal sonography when prolonged labor was diagnosed.
Time Frame: active labor
Population: Fetal head position was assessed successfully using transabdominal ultrasound in 142/150 women. Position could not be diagnosed in eight cases due to shadowing from maternal pelvis in cases at low stations.
Measure: Number; unit: percentage of participants in each group
Groups:
- Transabdominal Ultrasound: Fetal head position was assessed using a transabdominal scan
Arm/Group | Transabdominal Ultrasound
Number analyzed (Participants) | 142
percentage of participants in each group
  Cesarean section in cases with OP position (n=50) | 38
  Cesarean sin cases with non-OP position (n=92) | 17
Statistical Analysis 1: Comparison: Transabdominal Ultrasound; Test type: Superiority or Other; p = 0.01, Chi-squared

ADVERSE EVENTS:
Time Frame: Postpartum period
Groups:
- Transabdominal and Transperineal Sonography: Fetal head position was assessed using a transabdominal scan and fetal station was assessed by transperineal scan
Arm/Group | Transabdominal and Transperineal Sonography
Serious Adverse Events (participants affected / at risk) | 0/150
Other Adverse Events (participants affected / at risk) | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes